CLINICAL TRIAL: NCT06387810
Title: Irinotecan Liposome II in Combination With 5-FU/LV and Oxaliplatin in Perioperative Treatment of Borderline Resectable Pancreatic Cancer：A Prospective, Single-arm, Multicenter, Phase II Study
Brief Title: Irinotecan Liposome II in Combination With 5-FU/LV and Oxaliplatin in Perioperative Treatment of Borderline Resectable Pancreatic Cancer
Acronym: undetermined
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-PC-II-010
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-04

CONDITIONS: Borderline Resectable Pancreatic Cancer
Keywords: perioperative treatment, irinotecan liposome II
MeSH Terms: interventions — Oxaliplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined treatment group (Experimental): After screening and signing informed consent, patients who met the admission requirements received 4 cycles of neoadjuvant therapy with irinotecan liposome II combined with 5-FU/LV and oxaliplatin before surgery.
  Surgery was performed within 2 to 4 weeks after the end of neoadjuvant therapy. 4 to 6 weeks after surgery, 4 cycles of postoperative adjuvant therapy with irinotecan liposome II combined with 5-FU/LV and oxaliplatin was performed according to the investigator's judgment (once every 2 weeks, a 2-week cycle).
  Interventions: Drug: irinotecan liposome II combined with 5-FU/LV and oxaliplatin

INTERVENTIONS:
Drug: irinotecan liposome II combined with 5-FU/LV and oxaliplatin — irinotecan liposome II: 60mg/m2, intravenously for at least 90min, D1, administered every 2 weeks; oxaliplatin: 85 mg/m2, intravenous infusion, D1, every 2 weeks; calcium leucovorin: 400 mg/m2, 30±10min intravenously, D1, every 2 weeks; 5-fluorouracil: 2400 mg/m2 intravenously for 46-48 hours or according to study Center clinical practice, D1, administered every 2 weeks.
  Irinotecan liposome II, oxaliplatin, LV and 5-FU were given successively, and corresponding prophylactic administration could be selected according to clinical needs.
  Other Names: surgery

SUMMARY:
This is a prospective, single-arm, phase II study to evaluate the efficacy and safety of irinotecan liposome II in combination with oxaliplatin and 5-FU/LV in perioperative treatment of borderline resectable pancreatic cancer in 45 patients.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II study to evaluate the efficacy and safety of irinotecan liposome II in combination with oxaliplatin and 5-FU/LV in perioperative treatment of borderline resectable pancreatic cancer in 45 patients.

After screening and signing informed consent, patients who met the admission requirements received neoadjuvant therapy with irinotecan liposome II combined with 5-FU/LV and oxaliplatin before surgery (once every 2 weeks, every 2 weeks). After completing 4 cycles of preoperative neoadjuvant therapy, surgical evaluation was performed:

For patients evaluated for radical surgical resection, surgery was performed within 2 to 4 weeks after the end of neoadjuvant therapy, abdominal enhanced CT/MRI was performed within 4 to 6 weeks after surgery, and postoperative adjuvant therapy with irinotecan liposome II combined with 5-FU/LV and oxaliplatin was performed according to the investigator's judgment (once every 2 weeks, a 2-week cycle). After the completion of 4 cycles of postoperative adjuvant therapy, the tumor progression follow-up/survival follow-up stage was entered.

Patients who were assessed as not eligible for radical surgical resection could choose follow-up treatment according to the investigator's judgment, and continue to follow up their survival until withdrawal of informed consent or death.

ELIGIBILITY:
Inclusion Criteria:

* According to the NCCN Clinical Practice Guidelines for Pancreatic Cancer (2024.V1 edition), patients with critically resectable pancreatic cancer.
* Have at least one measurable lesion as a target lesion (according to RECIST v1.1);
* Have not received any anti-tumor therapy (including radiotherapy, ablation, chemotherapy, targeting, immunotherapy, etc.) or investigational drug therapy;
* ECOG: 0 ~ 1;
* Expected survival ≥3 months;
* Adequate organ and blood function

Exclusion Criteria:

* Pancreatic cancer of non-pancreatic ductal origin includes patients with pancreatic neuroendocrine carcinoma, pancreatic acinar cell carcinoma, pancreatic blastoma, and solid pseudopapillary tumor
* Severe gastrointestinal dysfunction
* Severe infection occurred within 4 weeks prior to initiation of treatment (CTCAE > Grade 2)
* Blood clotting is abnormal, has a tendency to bleed, or is receiving thrombolytic or anticoagulant therapy
* Have clinical symptoms or diseases of heart that are not well controlled, such as: (1) NYHA grade 2 or above heart failure; (2) Unstable angina pectoris; (3) Myocardial infarction occurred within 6 months; (4) Patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention
* Known allergy to irinotecan liposome II, other liposome products, oxaliplatin, 5-FU, calcium leucovorin, and any component of the above products
* Known peripheral neuropathy (CTCAE≥ Grade 3)
* In the investigator's judgment, subjects had other factors that might have led to their being forced to terminate the study, such as non-adherence to the protocol, other serious medical conditions (including mental illness) requiring combined treatment, clinically significant abnormalities in laboratory test values, or family or social factors that might affect subjects' safety or the collection of trial data

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
event free survival | 5 years
  The time between the date the subject started treatment and the occurrence of tumor progression leading to inoperability, postoperative recurrence/metastasis, or death, whichever occurred first.

SECONDARY OUTCOMES:
overall survival | 5 years
  The time from the start of treatment until death from any cause
R0 resection rate | 2 years
  R0 resection rate, defined as postoperative assessment of R0 resection (complete resection of the tumor, no cancer cells found on the margin of resection under the microscope, no cancer cells remaining under the naked eye or microscope, complete resection of the lesion). The proportion of subjects.
R1 excision rate | 2 years
  R1 excision rate, defined as postoperative assessment of R1 excision (microscopic residual, removal of all large lesions, submicroscopic margin of cancer). The proportion of subjects;
adverse event | 5 years
  Adverse events (AE)/Serious Adverse Events (SAE) (as determined by NCI-CTCAE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Wu, doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China